CLINICAL TRIAL: NCT07213622
Title: The Use of Smart Glasses for Saphenous Nerve Adductor Canal Block
Acronym: SMART
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Adam Zurney, Attending Anesthesiolgist, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000465
Record Dates: First submitted 2025-10-02; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Total Knee Arthroplasty
Keywords: Total knee arthroplasty
MeSH Terms: interventions — Smart Glasses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartglasses (Experimental)
  Interventions: Procedure: Smartglasses
- Standard of care (No Intervention)

INTERVENTIONS:
Procedure: Smartglasses — Wearing smart glasses while performing a nerve block
  Arms: Smartglasses

SUMMARY:
The use of smart glasses for saphenous nerve adductor canal blocks compared to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years or greater
* undergoing total knee arthroplasty

Exclusion Criteria:

* Patients with local infection at nerve block site
* BMI >40
* Patients who are at risk for local anesthesia systemic toxicity due to intraoperative local dose
* Patients with nerve damage to the femoral or saphenous nerve
* Documented history of mental or cognitive disabilities in EMR
* Non-English speaking patient
* Pregnant Women (self-reported)
* Prisoners
* Patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Time from needle insertion to complete local anesthetic injection | Until the end of the study

SECONDARY OUTCOMES:
Number of needle adjustments by user, ergonomics, head adjustments | until the end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- MetroHealth Hospital, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No